CLINICAL TRIAL: NCT05641415
Title: Finnish Imaging of Shoulder Study on the Prevalence of Imaging Findings of the Shoulder and Their Relevance to Clinical Symptoms in the General Population.
Brief Title: Finnish Imaging of Shoulder Study
Acronym: FIMAGE
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Simo Taimela, Adjunct Professor, University of Helsinki
Other Study IDs: HUS/13564/2022
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Pain; Rotator Cuff Tears; Glenoid Labrum Tear; Osteo Arthritis Shoulders
Keywords: Prevalence; Imaging; Shoulder; Clinical Examination; Asymptomatic; General population; Shoulder Function
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population sample: 600 participants aged 40 to 75 years will be randomly selected from a nationally representative general population sample of 9,922 individuals
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — MRI and x-ray of both shoulders

SUMMARY:
In the Finnish Imaging of Shoulder study we will recruit 600 participants from a nationally representative general population sample. Participants aged 40 to 75 years will be invited to a clinical visit that includes assessment of general health, shoulder history and symptoms, and bilateral clinical examination and shoulder imaging (both plain radiography and MRI). We aim to assess the prevalence of abnormal imaging findings in both asymptomatic and symptomatic individuals and explore possible risk factors for abnormal imaging findings and shoulder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Participation in the Health 2000 Survey
* Informed Consent

Exclusion Criteria:

* Dementia
* Terminal Cancer
* Previous shoulder joint replacement
* Contraindications for MRI

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population-based sample
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | At baseline
  Patient reported outcome measure.
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. A SPADI total score ranging from 0 (best) to 100 (worst) is produced by averaging the two subscale scores.
Constant -Murley Score | At baseline
  The Constant-Murley Score was designed to assess the functional state of a shoulder and contains both physician-completed and patient-reported portions. The four domains include pain (15 possible points), activities of daily living (20 possible points), mobility (40 possible points), and strength (25 possible points). Scores range from 0 points (most disability) to 100 points (least disability).

SECONDARY OUTCOMES:
Subjective Shoulder Value (SSV) | At baseline
  The SSV score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
Pain NRS | At baseline
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
EQ-5D-5L | At baseline
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.

OTHER OUTCOMES:
Shoulder Magnetic Resonance Imaging (MRI) | At baseline
  3T bilateral shoulder MRI
Shoulder Radiography | At baseline
  Plain radiographs (three projections) of both shoulders
Clinical Shoulder Examination | At baseline
  The clinical examination will include measurement of height, weight, active and passive range-of-motion (ROM) of both shoulders using an inclinometer and isometric muscle strength of shoulder abduction, internal, and external rotation. In addition, we will perform special shoulder tests following a structured assessment protocol
Hospital Anxiety and Depression Scale (HADS) | At baseline
  A self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic. Each item is answered by the patient on a four point (0-3) response category so the possible scores range from 0 to 21 for anxiety and 0 to 21 for depression (higher scores indicating a more severe disorder).
Pain Catastrophizing Scale (PCS) | At baseline
  The PCS was developed to help quantify an individual's pain experience, asking about how they feel and what they think about when they are in pain. The PCS asks 13 questions on thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. PCS total scores range from 0 - 52.
Pain Self Efficacy Questionnaire (PESQ) | At baseline
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain. High scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibounig T, Buchbinder R, Sillanpaa N, Ramo L, Toivonen P, Raatikainen S, Koskinen S, Harkanen T, Rissanen H, Czuba T, Paavola M, Jarvinen T, Taimela S; FIMAGE investigators. Concordance of shoulder symptoms and imaging findings: a protocol for the Finnish Imaging of Shoulder (FIMAGE) study. BMJ Open. 2023 Dec 28;13(12):e074457. doi: 10.1136/bmjopen-2023-074457. PMID 38154899